CLINICAL TRIAL: NCT03690687
Title: Delayed Small-Bowel Anastomosis in Patients With Postoperative Peritonitis Due to Nontraumatic Small-Bowel Perforation and Anastomotic Leak: Cohort Study
Brief Title: Delayed Small-Bowel Anastomosis in Patients With Postoperative Peritonitis
Acronym: Peritonitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Andrey Nikolayevich Zharikov (Other)
Responsible Party: Sponsor-Investigator, Andrey Nikolayevich Zharikov, Professor, Altai State Medical University
Organization: Altai State Medical University (Other)
Other Study IDs: Postoperative peritonitis
Record Dates: First submitted 2018-09-26; First posted 2018-10-01 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Postoperative Peritonitis; Anastomotic Leakage; Intestinal Perforation Small
Keywords: Surgical Anastomosis; Enterostomy; Mortality; Morbidity; Abdominal Closure Techniques; APACHE II; Secondary Peritonitis; Delayed Anastomosis; Primary Anastomosis; Mannheim Peritonitis Index
MeSH Terms: conditions — Anastomotic Leak; Peritonitis | interventions — Enterostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I. Primary anastomosis: Resection of the small bowel to place primary anastomosis into small intestine or transverse colon during relaparotomy.
  Interventions: Procedure: Primary anastomosis
- Group II. Delayed anastomosis: Resection of the small intestine to place delayed anastomosis. After the closure of the afferent and efferent loops of the small intestine, anastomosis was not applied. A decompression probe was introduced into the upper small intestine. In 24-36 hours, delayed anastomosis was placed into the small intestine or transverse colon during the planned relaparotomy with arrested postoperative peritonitis.
  Interventions: Procedure: Delayed anastomosis
- Group III. Enterostomy: Resection of the small intestine with enterostomy. In case there was no postoperative peritonitis relief and was organ dysfunction progression, anastomosis was not placed. The surgery was completed with enterostomy to perform open abdomen.
  Interventions: Procedure: Enterostomy

INTERVENTIONS:
Procedure: Primary anastomosis
  Groups: Group I. Primary anastomosis
Procedure: Delayed anastomosis
  Groups: Group II. Delayed anastomosis
Procedure: Enterostomy
  Groups: Group III. Enterostomy

SUMMARY:
Surgical management results for 114 patients with postoperative peritonitis due to small-bowel perforations, necrosis, and anastomotic leakage were comparatively analyzed. Using the APACHE-II (Acute Physiology, Age, Chronic Health Evaluation) and MPI (Mannheim Peritonitis Index) scoring systems, different surgical approaches were examined in three patient groups (primary anastomosis, delayed anastomosis, and enterostomy).

DETAILED DESCRIPTION:
One hundred and fourteen (114) participants with postoperative peritonitis resulted from small-bowel perforations or small-bowel anastomotic leaks were divided prior to surgery into 3 groups following the APACHE-II (Acute Physiology, Age, Chronic Health Evaluation) and MPI (Mannheim Peritonitis Index) scores, and different surgical approaches were applied to the groups: group I underwent resection of the small intestine to place primary anastomosis; group II was subjected to resection of the small intestine to place delayed anastomosis; and group III went through resection of the small intestine with enterostomy. The surgeon used minimization (including a random element) and stratification by gender, age, and small-bowel pathology.

The patients received resection of the small bowel to place primary small-bowel anastomosis, or as depending on their grouping:

* Resection of the small bowel to place primary anastomosis: resection of the small bowel to place primary anastomosis into small intestine or transverse colon were performed by routine practice during relaparotomy.
* Resection of the small intestine to place delayed anastomosis: resection of the small bowel was performed by routine practice. After the closure of the afferent and efferent loops of the small intestine, anastomosis was not applied. A decompression probe was introduced into the upper small intestine. In 24-36 hours, delayed anastomosis into small intestine or transverse colon was performed during the planned relaparotomy with arrested postoperative peritonitis.
* Resection of the small intestine with enterostomy: resection of the small intestine was performed by routine practice. In case there was no postoperative peritonitis relief and was organ dysfunction progression, anastomosis was not placed. The surgery was completed with enterostomy to perform open abdomen.

The specificity of each operation, including a decision to make changes in the planned anastomosis after assessing the severity of illness and the severity of postoperative peritonitis, was at the discretion of the surgeon.

All of the patients were followed up after operations. The patients were supervised in the clinic for 60 days post-surgery. During the postoperative period, complications in the three patient groups were assessed in terms of newly emerged small-bowel perforations, the number of anastomotic leaks, the number of programmed relaparotomies and on-demand relaparotomies, and mortality rate.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of postoperastive peritonitis
* Conducting relaparotomy

Exclusion Criteria:

* Peritoneal cancer
* Multiple organ dysfunction syndrome

Ages: 19 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Local patients admitted to the clinic from around Altai Krai cities, suffering from postoperative peritonitis due to small-bowel perforations and small-bowel anastomotic leaks
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with recurrent anastomotic leakage | up to 2 months
  Number of patients in groups 1 and 2

IPD SHARING:
Plan to Share IPD: No
The first group included 47 patients (41.2%) who underwent conventional surgical management during relaparotomy, taking into account APACHE-II severity of illness and MPI severity of peritonitis. This surgical treatment involved suturing the intestinal wall defects or small-bowel resection to place primary anastomosis. The second patient group included 55 patients (48.2%) to which the delayed anastomosis technique was applied during relaparotomy, taking account the APACHE-II and MPI scores. The third patient group included 12 patients (10.5%) who had the highest risk of small-bowel suture failure when closing the defects in either primary or delayed anastomosis, as well as the risk of new small-bowel perforations to occur. In these cases, resection of the intestine was performed with enterostomy, along with planned relaparotomies and Open Abdomen management.

REFERENCES:
- [Background] Zharikov AN, Lubyansky VG, Aliev AR. Surgical techniques for open abdomen in patients with postoperative peritonitis. Bulletin of Medical Science 2(10):76-80, 2018. URL: http://www.agmu.ru/files/%E2%84%962(10)2018.pdf
- [Background] Zharikov AN, Lubyansky VG, Aliev AR et al. Staged surgical treatment with temporary laparostomy in patients with postoperative peritonitis. Moscow Surgical Journal 1(41):10-14, 2015. URL: http://mossj.ru/journal/MOSSJ_2015/MXG_2015_01.pdf
- [Result] Zharikov AN, Lubyansky VG, Zharikov AA. A differentiated approach to repeat small-bowel anastomoses in patients with postoperative peritonitis: a prospective cohort study. Eur J Trauma Emerg Surg. 2020 Oct;46(5):1055-1061. doi: 10.1007/s00068-019-01084-7. Epub 2019 Feb 4. PMID 30719528